CLINICAL TRIAL: NCT03219060
Title: Motivational Interviewing as a Smoking Cessation Strategy With Nurses: an Exploratory Randomized Controlled Trial Following the MRC's Framework for Complex Interventions
Brief Title: Motivational Interviewing for Nurses' Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Government of Navarra (Unknown)
Responsible Party: Principal Investigator, Agurtzane Mujika, Dr. Agurtzane Mujika, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PENDING
Record Dates: First submitted 2017-07-10; First posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Health Behavior; Smoking Cessation; Health Personnel Attitude
Keywords: Cognitive dissonance; Motivational interviewing; Health Professional role; Nurses; Health Promotion; Lifestyle; Smoking cessation
MeSH Terms: conditions — Health Behavior; Smoking Cessation | interventions — Motivational Interviewing; Nurses; Crisis Intervention

ARMS (2):
- Intervention group (Experimental): MI based four individual sessions
  Interventions: Behavioral: Motivational interviewing for smoking cessation in nurses
- Control group (Active Comparator): Brief advice following 5As
  Interventions: Behavioral: Brief advice

INTERVENTIONS:
Behavioral: Motivational interviewing for smoking cessation in nurses — Intervention, four one-to-one sessions on an approximately weekly basis, with 3 components: MI context, toolkit, and relapse prevention. The sessions were embedded in a MI context and followed two phases: exploratory and resolutive. The former explored the potential ambivalence that nurses experienced and constructed motivation for change; the latter reinforced the decision to quit and developed a change plan. Participants could choose over a range of tools: some more helpful in the exploratory phase (i.e. decisional balance sheet) and others in the resolutive phase (i.e. problem solving skills). The third component was directed at maintenance strategies. The therapy stayed with the nurses in terms of where they were in relation to they readiness for change.
  Arms: Intervention group
Behavioral: Brief advice — Brief advice based on 5As
  Arms: Control group

SUMMARY:
This study's objective was to test the efficacy, acceptability and feasibility of a motivational interviewing (MI) based smoking cessation intervention with nurses.

DETAILED DESCRIPTION:
Despite the important role that health professionals have in reducing tobacco use, many have a smoking habit themselves. The prevalence of smoking is particularly high among nurses. A smoking cessation intervention for nurses who smoked, based on MI, was designed and evaluated following the UK Medical Research Council's (MRC) framework for complex interventions.

ELIGIBILITY:
Inclusion Criteria:

* Nurses who were smokers
* Nurses willing to participate in the study

Exclusion Criteria:

* Nurses who were pregnant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Biochemically verified smoking cessation | Following nurses' self-report of quitting (end of intervention (1 month) to 3 month follow-up)
  Urine sample collected in nurses who self-reported being abstinent for at least one week
Participant satisfaction | End of intervention (1 month)
  Client Satisfaction Questionnaire (CHQ-8) (Roberts et al 1984)
Duration of sessions | End of intervention (1 month)
  Following researcher's diary records

SECONDARY OUTCOMES:
Changes in Mean cigarettes smoked | Baseline, end of intervention (1 month) and 3 month follow-up
  Number of cigarettes smoked
Changes in Stages of change | Baseline, end of intervention (1 month) and 3 month follow-up
  Assessment of desire and readiness to quit smoking (Prochaska and Velicer, 1997)
Changes in Nicotine Dependence | Baseline, end of intervention (1 month) and 3 month follow-up
  Assessment of nicotine dependence using the Fagerström Test for Nicotine Dependence (FTND) (Becoña and Vazquez, 1998)
Changes in Self-efficacy | Baseline, end of intervention (1 month) and 3 month follow-up
  Assessment of general self-efficacy using GSE scale (Scholz et al, 2002)
Changes in Depression score | Baseline, end of intervention (1 month) and 3 month follow-up
  Depression screening using the Patient Health Questionnaire (PHQ-9) (Kroenke et al 2001)
Adherence to MI | End of intervention (1 month)
  Assessment of intervention fidelity and adherence to MI principles using Motivational Interviewing Treatment Integrity (MITI) Code (Moyers et al 2005)

CONTACTS AND LOCATIONS:
Overall Officials: Agurtzane Mujika, PhD, Principal Investigator — University of Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Background] Mujika A, Arantzamendi M, Lopez-Dicastillo O, Forbes A. Health professionals' personal behaviours hindering health promotion: A study of nurses who smoke. J Adv Nurs. 2017 Nov;73(11):2633-2641. doi: 10.1111/jan.13343. Epub 2017 Jun 21. PMID 28543954
- [Background] Duaso MJ, Bakhshi S, Mujika A, Purssell E, While AE. Nurses' smoking habits and their professional smoking cessation practices. A systematic review and meta-analysis. Int J Nurs Stud. 2017 Feb;67:3-11. doi: 10.1016/j.ijnurstu.2016.10.011. Epub 2016 Nov 2. PMID 27880873
- [Background] Duaso MJ, McDermott MS, Mujika A, Purssell E, While A. Do doctors' smoking habits influence their smoking cessation practices? A systematic review and meta-analysis. Addiction. 2014 Nov;109(11):1811-23. doi: 10.1111/add.12680. Epub 2014 Aug 5. PMID 25041084
- [Result] Mujika A, Forbes A, Canga N, de Irala J, Serrano I, Gasco P, Edwards M. Motivational interviewing as a smoking cessation strategy with nurses: an exploratory randomised controlled trial. Int J Nurs Stud. 2014 Aug;51(8):1074-82. doi: 10.1016/j.ijnurstu.2013.12.001. Epub 2013 Dec 15. PMID 24433609